CLINICAL TRIAL: NCT02783820
Title: A Single Centre, Two-part, Phase I Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile of Ascending Oral Doses of MMV390048 and Its Antimalarial Activity Against Plasmodium Falciparum in Healthy Adult Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic Profile of Ascending Oral Doses of MMV390048, Part A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Clinical Network Services (CNS) Pty Ltd (Industry); Q-Pharm Pty Limited (Industry); QIMR Berghofer Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMV_MMV390048_16_01
Record Dates: First submitted 2016-05-19; First posted 2016-05-26 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Malaria
Keywords: malaria, single ascending dose,
MeSH Terms: conditions — Malaria | interventions — MMV390048

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- MMV390048 40 mg (Experimental): MMV390048 40 mg, tablets, single dose
  Interventions: Drug: MMV390048 40 mg
- Placebo to match MMV390048 40 mg (Placebo Comparator): Placebo to match MMV390048 40 mg, tablets, single dose
  Interventions: Drug: Placebo to match MMV390048 40 mg
- MMV390048 80 mg (Experimental): MMV390048 80 mg, tablets, single dose
  Interventions: Drug: MMV390048 80 mg
- Placebo to match MMV390048 80 mg (Placebo Comparator): Placebo to match MMV390048 80 mg, tablets, single dose
  Interventions: Drug: Placebo to match MMV390048 80 mg
- MMV390048 120 mg (Experimental): MMV390048 120 mg, tablets, single dose
  Interventions: Drug: MMV390048 120 mg
- Placebo to match MMV390048 120 mg (Placebo Comparator): Placebo to match MMV390048 120 mg, tablets, single dose
  Interventions: Drug: Placebo to match MMV390048 120 mg

INTERVENTIONS:
Drug: MMV390048 40 mg
  Arms: MMV390048 40 mg
Drug: Placebo to match MMV390048 40 mg
  Arms: Placebo to match MMV390048 40 mg
Drug: MMV390048 80 mg
  Arms: MMV390048 80 mg
Drug: Placebo to match MMV390048 80 mg
  Arms: Placebo to match MMV390048 80 mg
Drug: MMV390048 120 mg
  Arms: MMV390048 120 mg
Drug: Placebo to match MMV390048 120 mg
  Arms: Placebo to match MMV390048 120 mg

SUMMARY:
This Phase I study will evaluate the safety, tolerability and pharmacokinetic properties of escalating single doses of reformulated MMV390048 when administered to healthy men and women of non-childbearing potential (WNCBP) under fasted conditions (Part A).

DETAILED DESCRIPTION:
This Phase I study will evaluate the safety, tolerability and pharmacokinetic properties of escalating single doses of reformulated MMV390048 when administered to healthy men and women of non-childbearing potential (WNCBP) under fasted conditions (Part A).

Primary objectives:

• To evaluate the safety and tolerability of single ascending doses of MMV390048 administered orally to healthy subjects (men and WNCBP) under fasted conditions

Secondary objectives:

• To describe the pharmacokinetics of MMV390048 in healthy subjects (men and WNCBP) after single oral dose administration

ELIGIBILITY:
Inclusion Criteria:

1. Completion of the written informed consent process.
2. Men or WNCBP age 18 to 55 years, in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
3. Male subjects agree to use acceptable methods of contraception if the male subject's partner could become pregnant from the time of the first administration of study medication until 130 (90+40) days following administration of the investigational medicinal product. One of the following acceptable methods of contraception must be utilized:

   * Condom and occlusive cap (diaphragm or cervical/vault caps)
   * Surgical sterilization (vasectomy with documentation of azoospermia) and a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps].
   * The subject's female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps].
   * The subject's female partner uses medically prescribed topically-applied transdermal contraceptive patch and a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps].
   * The subject's female partner has undergone documented tubal ligation (female sterilization). In addition, a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps].
   * The subject's female partner has undergone documented placement of an intrauterine device or intrauterine system. In addition, a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps].
   * True abstinence: when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Abstinent subjects have to agree to use 1 of the above-mentioned contraceptive methods, if they start sexual relationships during the study and for up to 100 days after the last dose of study drug.
4. Women subjects must be of non-childbearing potential (WNCBP) as per one of the following definitions:

   * Natural (spontaneous) post-menopausal defined as being amenorrhoeic for at least 12 months without an alternative medical cause with a screening follicle stimulating hormone level consistent with local laboratory levels for post-menopause.
   * Premenopausal with irreversible surgical sterilization by hysterectomy and/or bilateral oophorectomy or salpingectomy at least 6 months before screening (as determined by subject medical history).
5. Haematology, clinical chemistry and urinalysis results at screening that are within the local laboratory reference range or, if outside the range, not clinically significant as judged by the Investigator. More specifically, serum creatinine, hepatic transaminase enzymes (AST ALT), and total bilirubin (unless the subject has documented Gilbert syndrome) should not exceed the upper laboratory norm and haemoglobin must be equal to or higher than the lower limit of the normal range.
6. Total body weight greater than 50 kg and a body mass index (BMI) within the range of 18 to 32 kg/m2 (inclusive).
7. Non-smoker or ex-smoker for more than 90 days prior to screening, or smoke no more than 5 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.
8. Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
9. Agree to stay in contact with the study site for the duration of the study and up to 2 weeks following the end of study visit, provide updated contact information as necessary, and have no current plans to move away from the study area for the duration of the study.

Exclusion Criteria:

1. Male subjects with a female partner(s) who is (are) pregnant or lactating from the time of the administration of study medication.
2. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means.
3. Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal (including gallbladder), cardiovascular (including a family history of long QT syndrome or sudden death), hepatic, psychiatric, neurologic, or allergic disease (including drug or food allergies, anaphylaxis or other severe allergic reactions but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
4. History of malignancy of any organ system (other than localised basal cell carcinoma of the skin), treated or untreated, within the past five years, regardless of whether there is evidence of local recurrence or metastases.
5. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
6. Any surgical or medical condition possibly affecting drug absorption (e.g. cholecystectomy, gastrectomy, bowel disease, etc.), distribution, metabolism or excretion.
7. Previous splenectomy.
8. A history of photosensitivity.
9. Subject positive for any of the following

   * Anti-human immunodeficiency virus 1 or 2 antibodies (anti-HIV1 or anti-HIV2 Ab) (ELISA)
   * Hepatitis B surface antigen (HBsAg)
   * Anti-hepatitis B core antibodies (anti-HBcAb)
   * Anti-hepatitis C antibodies (anti-HCV)
10. Resting vital signs (measured after 5 minutes in the supine position) at screening, pre-dose (Part A) or pre-inoculation (Part B) outside of the following study-specific normal ranges:

    * tympanic body temperature < 38.0 °C
    * 90 < SBP < 140 mmHg
    * 50 < DBP < 90 mmHg
    * 40 < pulse rate < 100 bpm
11. Symptomatic postural hypotension at screening, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg 2 minutes after changing from a supine to standing position.
12. A history of clinically significant ECG abnormalities, or any of the following ECG abnormalities at screening, pre-dose (Part A and B) or pre-inoculation (Part B):

    * PR >210 ms
    * QRS complex >120 ms
    * QTcF >450 ms
    * Second or third degree atrioventricular block
    * Incomplete, complete or intermittent bundle branch block
    * Abnormal T wave morphology
    * Left ventricular hypertrophy with repolarisation abnormalities
    * Right ventricular hypertrophy.
13. Presence of acute infectious disease or fever (i.e. tympanic body temperature ≥38.5 ºC) within five days prior to the first dose of study medication (Part A) or the inoculation administration (Part B).
14. Use of prescription or non-prescription drugs, herbal and dietary supplements within 14 days or 5 half-lives (whichever is the longer) prior to the first dose of study medication (Part A) or the inoculation administration (Part B). [As an exception, paracetamol may be used at doses of up to 1 g/day (Part A) or 2 g/day (Part B), or ibuprofen up to 1.2 g/day (Part B). Limited use of other non-prescription medications not believed to affect subject safety or the overall results of the study, may be permitted on a case-by-case basis following approval by the sponsor.]
15. Recipient of any vaccination within 28 days prior to the first dose of study medication (Part A) or the inoculation administration (Part B).
16. Urine drug screen at screening, pre-dose (Part A) or pre-inoculation (Part B) positive for any drug as listed in Section 9.2.4 unless there is an explanation acceptable to the medical Investigator (e.g. the subject has stated in advance that they consumed a prescription or over the counter product which contained the detected drug) and/or the subject has a negative urine drug screen on retest by the pathology laboratory.
17. Ingestion of any poppy seeds within the 24 hours prior to the screening blood test.
18. A positive alcohol breath test at screening, pre-dose (Part A) or pre-inoculation (Part B).
19. History of regular alcohol consumption exceeding a weekly intake of more than 21 units for males and more than 14 units for females (one unit is equivalent to 8-10 g of ethanol, 285 ml of beer or lager, one glass [125 ml] of wine, or 25 ml of spirits) within 6 months of screening.
20. History of drug habituation, or any prior intravenous usage of an illicit substance.
21. Participation in any investigational product study within 12 weeks or five half-lives (whichever is longer) prior to the first dose of the study medication.
22. Intake of grapefruit, grapefruit juice or grapefruit-related citrus fruits (e.g. Seville oranges, pomelos) within 28 days prior to the first dose of the study medication.
23. Excessive consumption of beverages containing xanthine bases (e.g. more than 400 mg of caffeine per day, equivalent to approximately 4 cups of coffee).
24. Pregnant or nursing (lactating) women.
25. Participation in any research study involving blood sampling (more than 450 ml/ unit of blood), or blood donation to the Australian Red Cross Blood Service (ARCBS) or other blood bank during the 8 weeks prior to IMP administration (Part A) or inoculation (Part B).
26. Blood donation (excluding plasma donation) of any volume, within 1 month prior to screening.
27. Medical requirement for intravenous immunoglobulin or blood transfusions.
28. Subject with poor peripheral venous access.
29. Subject unwilling or unable to comply with the restrictions described in this protocol.
30. Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
31. Any subject who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
32. Recent (within the last three years) and/or recurrent history of autonomic dysfunction (e.g. recurrent episodes of fainting, palpitations, etc.).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, Prof, Principal Investigator — Q-Pharm Pty Ltd and QIMR Berghofer Medical Research Institute
Locations (1):
- Q Pharm Clinics, Herston, Australia

IPD SHARING:
Plan to Share IPD: Yes
Clinical safety data (physical exam, ECG, vital signs, clinical score, AEs) lab safety data PK data PCR data Dosing completed, subject withdrawals,significant protocol deviations. Serious Adverse Event Reports

REFERENCES:
- [Derived] McCarthy JS, Donini C, Chalon S, Woodford J, Marquart L, Collins KA, Rozenberg FD, Fidock DA, Cherkaoui-Rbati MH, Gobeau N, Mohrle JJ. A Phase 1, Placebo-controlled, Randomized, Single Ascending Dose Study and a Volunteer Infection Study to Characterize the Safety, Pharmacokinetics, and Antimalarial Activity of the Plasmodium Phosphatidylinositol 4-Kinase Inhibitor MMV390048. Clin Infect Dis. 2020 Dec 17;71(10):e657-e664. doi: 10.1093/cid/ciaa368. PMID 32239164

RESULTS

PARTICIPANT FLOW:
Groups:
- Pooled Placebo: Pooled placebo from all cohorts (2 per cohort = 6)
Period: Overall Study
Arm/Group | Pooled Placebo | MMV390048 40 mg | MMV390048 80 mg | MMV390048 120 mg
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | MMV390048 40 mg | MMV390048 80 mg | MMV390048 120 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (11.3) | 24.8 (2.5) | 23 (2.6) | 40.2 (13.9) | 30.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 5 | 5 | 2 | 5 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.1 (2.4) | 23.4 (1.9) | 24.3 (3.2) | 25.4 (3) | 24.3 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Safety of MMV390048 - Number of Adverse Events
Description: Number of observed and self-reported Adverse Events (AE) (unexpected toxicities, adverse events encountered during or after investigational drug administration)
Time Frame: 28 days post administration of a single oral dose of MMV390048 to healthy volunteers
Measure: Number; unit: Number of adverse events
Arm/Group | Pooled Placebo | MMV390048 40 mg | MMV390048 80 mg | MMV390048 120 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Number of adverse events | 13 | 0 | 9 | 12

2. Secondary Outcome: PK Cmax
Description: Estimation of the maximum plasma concentration over 28 days post administration of a single dose of MMV390048 using non-compartmental methods
Time Frame: 28 days
Reporting Status: Not Posted

3. Secondary Outcome: PK Tmax
Description: Estimation of the time to maximum plasma concentration over 28 days post administration of a single dose of MMV390048 using non-compartmental methods
Time Frame: 28 days
Reporting Status: Not Posted

4. Secondary Outcome: PK Total Exposure AUClast
Description: Estimation of the last quantifiable concentration over 28 days post administration of a single dose of MMV390048 using non-compartmental methods
Time Frame: 28 days
Reporting Status: Not Posted

5. Secondary Outcome: PK Total Exposure AUCinf
Description: Estimation of the area under the plasma concentration time curve over 28 days post administration of a single dose of MMV390048 using non-compartmental methods
Time Frame: 28 days
Reporting Status: Not Posted

6. Secondary Outcome: PK Distribution and Clearance (CL/F)
Description: Apparent oral clearance (CL/F) over 28 days post administration of a single dose of MMV390048 using non-compartmental methods
Time Frame: 28 days
Reporting Status: Not Posted

7. Secondary Outcome: PK Distribution and Clearance (Vz/F)
Description: Apparent volume of distribution (Vz/F) over 28 days post administration of a single dose of MMV390048 using non-compartmental methods
Time Frame: 28 days
Reporting Status: Not Posted

8. Secondary Outcome: PK Distribution and Clearance (t½)
Description: Terminal half-life (t½) over 28 days post administration of a single dose of MMV390048 using non-compartmental methods
Time Frame: 28 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Until Day 28
Arm/Group | Pooled Placebo | MMV390048 40 mg | MMV390048 80 mg | MMV390048 120 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 0/6 | 4/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=6) | MMV390048 40 mg (N=6) | MMV390048 80 mg (N=6) | MMV390048 120 mg (N=6)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=6) | MMV390048 40 mg (N=6) | MMV390048 80 mg (N=6) | MMV390048 120 mg (N=6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site reaction (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 4 (5)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sterile pyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suture insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days